CLINICAL TRIAL: NCT06857734
Title: The Analgesic and Anti-inflamatory Effect of Vitamin B Versus Vitamin C Infusion in Patients Undergoing Laparoscopic Cholecystectomy ; a Randomized Controlled Trial
Brief Title: Analgesic and Anti-inflamatory Effect of Vit. B
Acronym: vit B/vit C
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Islam Moawad, Resident, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ms 33-12-2024
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Vitamin B Complex; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group B (Experimental)
  Interventions: Drug: Vitamin B Complex
- Group C (Experimental)
  Interventions: Drug: vitamin C
- Group N (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin B Complex — group of vit. B will recieve as an oral capsules for 4 days preoperative , and infusion of vitamin B complex 1ml diluted in 100 ml normal saline administered intravenously after anathesia induction .
  Arms: Group B
Drug: vitamin C — group of vitamin C will recieve 1000 mg as an oral capsule for 4 days and infusion at dose of 50 mg/kg diluted in 100 ml normal saline administered iv after induction of anathesia .
  Arms: Group C
Drug: Placebo — patients will recieve placebo tablets with identical regimen preoperative and a placebo infusion of 100 ml normal saline after induction of anathesia ,prepared with identical appearance and taste by the pharmacist according to the randomization group.
  Arms: Group N

SUMMARY:
Vitamin C, also known as ascorbic acid, is a potent reducing agent and antioxidant that plays a crucial role in various metabolic processes.Vitamin B complex, a group of eight essential B vitamins, plays a crucial role in cellular metabolism, energy production, and maintaining nervous system health. There are few available studies on the effects of vitamin B injection on plasma inflammatory markers and its adjuvant analgesic effect along with the routine multimodal analgesia. Considering limited research and existing controversies in this field, the aim of present study is to evaluate the effects of preoperative and intraoperative vitamin B12 administration compared to vitamin C when used as a component of the multimodal analgesic technique in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-60 years)
* American Society of Anesthesiologists (ASA) classification I-II
* Patients undergoing laparoscopic cholecystectomy under general anaesthesia

Exclusion Criteria:

* Hypersensitivity to vitamin B complex or vitamin C
* History of chronic pain or use of opioids within the last month
* Patient with inflammatory conditions
* Severe renal or hepatic impairment
* Patient with intellectual disabilities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The total dose of analgesics required postoperatively | within the first 24 hours and the time to first request

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes